CLINICAL TRIAL: NCT00884702
Title: Regional Rates of Cerebral Protein Synthesis: Effects of Sleep and Memory Consolidation
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090123; 09-M-0123
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04-18

CONDITIONS: Brain Mapping
Keywords: Sleep; 14C-Leucine; Cerebral Protein Synthesis; Memory; Positron Emission Tomography (PET); HV; Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* The brain needs sleep to function normally, but the purpose of sleep is not understood. Brain activity decreases during sleep, so it may be that sleep is important to maintain, repair, or reorganize brain cells. In animals, the formation of brain proteins increases during sleep, and the same thing may happen in humans.
* There is also evidence that learning and memory are helped by sleep, and that the synthesis of proteins in the brain are involved.

Objectives:

* To examine the formation of proteins in the brain while people are awake, deprived of sleep, and during sleep.
* To look at the formation of proteins in the brain while awake or asleep and following learning a task.

Eligibility:

* Healthy volunteers between 18 and 28 years of age.
* Volunteers must not have psychiatric, neurologic, or sleep disorders or certain types of vision problems, and must be able to undergo imaging studies.

Design:

* Study Part I (protein formation in waking, sleep deprivation, and sleep):
* Participants will wear an actigraph (a unit to record motor activity) for 2 weeks prior to admission.
* Participants will have physical and psychological examinations, along with a blood sample.
* After admission participants will have three positron emission tomography (PET) scans to study protein formation and one magnetic resonance imaging (MRI) scan over the course of two days.
* Participants may be asked to stay awake for as long as 20 hours and will be monitored throughout.
* Participants will be able to sleep overnight after they complete the required scans and monitoring, and will be discharged the following morning.
* Study Part II (protein formation in waking and sleep combined with a learning task):
* Participants will wear an actigraph (a unit to record motor activity) for 2 weeks prior to admission.
* Participants will have physical and psychological examinations, along with a blood sample.
* After admission participants may be asked to stay awake for as long as 20 hours and will be monitored throughout.
* The next morning, participants will be trained to perform a computerized visual discrimination task, and will be tested 8 hours later (after sleep or after remaining awake) on the visual discrimination task.
* Some participants may have PET and MRI scans as part of the study.
* Participants will be able to sleep overnight after they complete the required tests and scans, and will be discharged the following morning.
* Participants will receive financial compensation for their participation in these studies.

DETAILED DESCRIPTION:
The importance of sleep is widely appreciated, but the actual function of sleep remains unknown. Sleep occurs in much of the animal kingdom, in all mammals and birds and even in some lower forms. Sleep deprivation impairs brain function, and in rats, total sleep deprivation for 2-3 weeks results in death. One hypothesized role of sleep is for restoration and reorganization of neuronal circuits. There is some indirect evidence that during sleep, when cerebral energy requirements are reduced, cell resources are diverted to protein synthesis for the restoration of structure and function. The objectives of the present study are: 1) to further define the relationship between regional rates of cerebral protein synthesis (rCPS) and sleep and 2) to ascertain whether sleep-dependent visual learning during slow wave sleep (SWS) results in increases in rCPS in the primary visual cortex. We propose to use a novel positron emission tomography (PET)-based technique to quantify regional rates of cerebral protein synthesis (rCPS) in young, adult, healthy volunteers. The first objective will be addressed in Part I in which we will study each subject under the following three conditions: 1) awake and sleep-sated, 2) awake and sleep-deprived, and 3) during SWS after sleep-deprivation. Our aim is to complete fully successful studies in 15 subjects. The second objective will be addressed in Part II in which we will assess the relationship between rCPS and sleep-dependent visual learning on a retinotopically specific task. Each participant will serve as his own control by comparing the trained primary visual cortex hemisphere with the untrained hemisphere to which comparable visual information is presented but without learning. In Part II we will study two groups of subjects: 1) One group will be studied during SWS following the training session; 2) The second group will be studied at the same interval following the training session but awake. Subjects will be monitored with polysomnography to identify the stages of sleep. Our aim in part II is to complete fully successful studies in 15 subjects in each of the two groups. We anticipate that the results of Part I will identify changes in rCPS in specific brain regions which are characteristic of SWS and results of Part II may reveal relationships between rCPS and memory consolidation during SWS.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy male and female volunteers who have no present or past diagnosis of neurologic, medical or psychiatric conditions which may confound either learning trails, normal sleep patterns or the ability to undergo sleep deprivation.

Healthy male and female subjects, 18-28 years of age, who do not meet any exclusion criteria, with self-reported normal sleep patterns (i.e., 6-9 h per night) and no major sleep disruptions during the four weeks prior to evaluation will be considered for inclusion in the study.

EXCLUSION CRITERIA INCLUDE A HISTORY OF, OR CURRENT:

1. chronic medical condition which is a contraindication for PET or MRI scanning,
2. past or present diagnosis of psychiatric conditions (DSM-IV criteria) (many conditions (e.g. depression), may confound performance on learning trails or be associated with baseline sleep abnormalities),
3. chronic/degenerative/acquired neurologic disorder, (4) family history of genetically transmissible neurologic disorder,

(5) sleep disorders or medical conditions associated with chronically disordered sleep which may confound performance on learning trails or interfere with the sleep requirements of this study,

(6) visual impairments which may confound performance on learning trails,

(7) claustrophobic subjects,

(8) subjects who meet the above inclusion criteria, but are unable to cooperate with the requirements of the study (e.g. refusal to wear actigraphs or maintain 10 hours time in bed, reported difficulty sleeping away from home or on their backs).

(9) Subjects with chronic indicated or non-indicated use of any medications which interfere with sleep architecture and/or learning trails will be excluded. Generally, we will prohibit the use of medications/agents (e.g. anti-histamines, benadryl, melatonin, cigarettes, chocolate, coffee, tea, caffeine drinks etc.), which have significant CNS penetration, are alerting, and/or disrupt physiologic sleep-wake cycles or sleep architecture, for the 72 hrs immediately preceding presentation for the study. To acclimatize subjects, we will encourage patients to discontinue or minimize the use of these agents/medications (e.g. less than or equal to 1 cup of coffee/day) at the time of initial screening (at the same time as actigraphy application, approximately 2 wks prior to the study).

Similarly, we ask subjects to minimize alcohol use for the 2 wks prior to the study and will discontinue alcohol use for the 72 hrs immediately preceding the study.

(10) Subjects who have used illicit drugs (marijuana, cocaine, heroin, etc.) within the immediate 2 wks preceding the study.

(11) Female subjects will be excluded if either clinical history is suspicious for, or laboratory evaluation is consistent with pregnancy.

(12) Subjects unwilling to undergo HIV testing, unless enrolling in Part IIa of the study.

(13) Subjects who test HIV positive.

(14) Patients with para- and/or ferro-magnetic prosthesis/implants/fragments in their body will be excluded from the study.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 538 (Actual)
Dates: Start 2009-04-16; Study Completion 2017-04-18

PRIMARY OUTCOMES:
Regional rates of cerebral protein synthesis | 48 hrs

SECONDARY OUTCOMES:
Sleep state and performance on visual discrimination task. | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn B Smith, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armitage R. Microarchitectural findings in sleep EEG in depression: diagnostic implications. Biol Psychiatry. 1995 Jan 15;37(2):72-84. doi: 10.1016/0006-3223(94)00082-E. PMID 7718683
- [Background] Bishu S, Schmidt KC, Burlin T, Channing M, Conant S, Huang T, Liu ZH, Qin M, Unterman A, Xia Z, Zametkin A, Herscovitch P, Smith CB. Regional rates of cerebral protein synthesis measured with L-[1-11C]leucine and PET in conscious, young adult men: normal values, variability, and reproducibility. J Cereb Blood Flow Metab. 2008 Aug;28(8):1502-13. doi: 10.1038/jcbfm.2008.43. Epub 2008 May 21. PMID 18493259
- [Background] Boyle PJ, Scott JC, Krentz AJ, Nagy RJ, Comstock E, Hoffman C. Diminished brain glucose metabolism is a significant determinant for falling rates of systemic glucose utilization during sleep in normal humans. J Clin Invest. 1994 Feb;93(2):529-35. doi: 10.1172/JCI117003. PMID 8113391
- [Derived] McWhirter KK, Morrow AS, Lee BA, Bishu S, Zametkin AJ, Balkin TJ, Smith CB, Picchioni D. A PILOT STUDY ON THE ENCODING OF A PERCEPTUAL LEARNING TASK FOLLOWING SLEEP DEPRIVATION. Percept Mot Skills. 2015 Aug;121(1):80-93. doi: 10.2466/23.PMS.121c11x9. Epub 2015 Jul 30. PMID 26226287